CLINICAL TRIAL: NCT03550235
Title: Exploration of Dyspnea at Non-high BNP
Brief Title: Exploration of Dyspnea at Non-high Brain Natriuretic Peptide (BNP)
Acronym: NEON HFpEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01621-52
Record Dates: First submitted 2018-04-27; First posted 2018-06-08 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart failure; dyspnea; stress test
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with unexplained stress dyspnea ( ≥ stage 2 NYHA), no significant underlying lung disease, with an ejection fraction > 50%, normal resting filling pressures, NTproBNP < 220 pg/ml in < 75 years, and < 450 pg/ml in ≥ 75 years will be studied with stress echocardiography and cardiometabolic stress test (VO2). These patients may have abnormal adaptation during exercise, suggesting that chronic symptoms may be related to a heart failure with preserved ejection fraction (HFPEF). More accurate and earlier diagnosis of HFPEF using stress echocardiography and VO2 may better manage stress dyspnea in patients and prevent progression of HFPEF.

A clinical assessment will be offered to people with unexplained stress dyspnea. The procedures and products used in this study are usually used as part of HFpEF's diagnostic strategy. During this assessment, carried out on an outpatient basis, an anamnesis collection, a cardiovascular clinical examination, an evaluation of dyspnea by the NYHA functional class and by 2 questionnaires, an electrocardiogram will be carried out, a 6-minute walk test, a biological blood test, a trans thoracic rest and stress cardiac ultrasound, respiratory functional tests (with diffusion capacity of lung for carbon monoxide (DLCO) and blood gas), and a metabolic stress test. A follow-up at 1 and 2 years is planned (visit, sampling and resting echocardiography).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 40 years of age, and under 80 years of age with unexplained effort dyspnea, able to pedal.
* Echocardiographic ejection fraction > 50%
* NTproBNP < 220 pg/ml in < 75 years, and < 450 pg/ml in ≥ 75 years

Exclusion Criteria:

* Patient with coronary, valve, hypertrophic, hypertensive, infiltrative, constrictive, or rhythmic, significant and/or progressive heart disease.

BMI > 35 kg/m².

* Unstable patient (systolic blood pressure < 90 mmHg, resting pulse > 100 BPM) or clinically congested (edema of the lower limbs, crackling in the lungs).
* Patient with Pulmonary function testing (EFR) showing significant respiratory disease (FEV1/ vital capacity (CV) max < 0.7, total lung capacities (CPT)< LIN)
* Chronic renal failure with creatinine clearance < 30 ml/min (MDRD) or dialysis
* Patient with anemia (Hb < 12 g/dl)
* Patient with hypo or hyperthyroidism on thyreostimulating hormone (TSH) value
* Patient under justice safeguard measure or guardianship

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All referred patients for unexplained dyspnea that must be assessed
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Occurence of HFpEF | during the 2 years of follow-up
  HFpEF diagnosis will be made in attendance of following symptoms:
  * heart failure
  * NTproBNP>125pg/ml
  * preservation of ejection fraction with Left Ventricular Ejection Fraction (LVEF)>50%
  * structural heart disease with expansion of left ventricular mass (VM) (men: VM≥115 g/m² or women ≥ 95 g/m² and an E/e' ratio≥13
dyspnea on exertion | during the 2 years of follow-up
NTproBNP levels at rest | during the 2 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle BERTHELOT, Dr, Principal Investigator — AP-HP Hôpital Bicêtre
Locations (4):
- France (4):
  - Hopital Bicêtre, Le Kremlin-Bicêtre
  - Polyclinique de Poitiers, Poitiers
  - CHU Pontchaillou, Rennes
  - CCM RANGUEIL - LARREY CHU toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No